CLINICAL TRIAL: NCT07364877
Title: A Randomized, Open-label, Single-dose, 2-sequence, Two-period, Crossover Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of DW4421 and DW4421S in Healthy Adult Volunteers
Brief Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetics of DW4421 and DW4421S in Healthy Adult Volunteers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW4421-104
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): cross-over
  Interventions: Drug: DW4421; Drug: DW4421S
- Sequence B (Experimental): Cross-over
  Interventions: Drug: DW4421; Drug: DW4421S

INTERVENTIONS:
Drug: DW4421 — DW4421 or DW4421S
Drug: DW4421S — DW4421 or DW4421S

SUMMARY:
Safety and pharmacokinetic characteristics evaluation of DW4421 and DW4421S

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 19 to 50 (inclusive) years
* Subjects weighing between 50 kg and 90 kg with BMI between 18 and 27 kg/m2 (inclusive)

Exclusion Criteria:

* clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 48 hour
AUC0-t | up to 48 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea